CLINICAL TRIAL: NCT03131570
Title: Safety and Efficacy of Secukinumab in Adults With Chronic Plaque Type Psoriasis With a PASI Score of 6 to 12
Brief Title: Safety and Efficacy of Secukinumab in Mild Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James G. Krueger, MD, PhD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, James G. Krueger, MD, PhD, Head of the Laboratory for Investigative Dermatology, Rockefeller University
Organization: Rockefeller University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKR-0937
Record Dates: First submitted 2017-03-10; First posted 2017-04-27 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Chronic Plaque Psoriasis; Secukinumab
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: To compare the secukinumab-receiving mild psoriasis subjects (Group 1) and the placebo-receiving mild psoriasis subjects (Group 2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 6 months of Secukinumab at a dose of 300 mg with injections administered once weekly at baseline and at weeks 1, 2, 3, and 4 and then every 4 weeks for 6 months of period.
  Interventions: Drug: Secukinumab
- Group 2 (Placebo Comparator): Placebo followed by Secukinumab. 3 months of placebo followed by 3 months of Secukinumab at a dose of 300 mg with injections administered once weekly at week 12 and at weeks 13, 14, 15, and 16 and then every 4 weeks for 3 months of period.
  Interventions: Drug: Placebo followed by Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Arms: Group 1 - Group 1 will receive Secukinumab at a dose of 300 mg with injections administered once weekly at baseline and at weeks 1, 2, 3, and 4 and then every 4 weeks for 6 months of period. In order to maintain the blind for the Group 2, Group 1 will receive placebo injections at weeks 13, 14, and 15. Group 1 will discontinue Secukinumab after 6 months of period being observed from week 25 to week 72 (48 weeks).
  Other Names: COSENTYX
  Arms: Group 1
Drug: Placebo followed by Secukinumab — Arms: Group 2 - Group 2 will receive placebo injections corresponding to the Group 1 regimen until week 8 in order to maintain a double-dummy design until week 12. From week 12, Group 2 will receive Secukinumab with injections administered once weekly at week 12 and at weeks 13, 14, 15, and 16 and then every 4 weeks for 3 months of period. Group 2 will discontinue Secukinumab after 6 months of period being observed from week 25 to week 72 (48 weeks).
  Other Names: Placebo followed by COSENTYX
  Arms: Group 2

SUMMARY:
Mild psoriasis not only progresses to moderate-to-severe psoriasis but also precedes systemic inflammation that leads to psoriatic arthritis and cardiovascular comorbidities. By curing mild psoriasis with a short-term anti- interleukin (IL)-17A treatment, investigators may reduce the costs of treating psoriasis and associated medical conditions, including psoriatic arthritis, cardiovascular disease, and diabetes.

DETAILED DESCRIPTION:
Psoriasis is an immune-mediated disease of the skin that, even in mild disease, increases the risk of comorbidities such as cardiovascular disease and metabolic derangements. Mild psoriasis tends to be treated with topical drugs, while moderate-to-severe disease is optimally treated with systemic immune modulators. However, the treatment of "mild" psoriasis needs to be re-thought because recent studies have revealed that mild psoriasis is characterized by stronger expression of pathogenic molecules, such as interleukin (IL)-17A, and higher numbers of T cells in the skin, compared to severe psoriasis. A key distinction between mild and severe psoriasis is now discovered to be the higher expression of negative immune regulatory genes in mild lesions. Therefore, targeted immune therapy with anti-IL-17A, which is highly effective in severe psoriasis, might be equally (or even more) effective in mild disease. Also, restoration of immune tolerance might be more easily achieved in mild disease. Thus, short-term anti-IL-17A treatment of mild psoriasis might prevent the recurrence and eventually cure the disease. The aim of study is to test this hypothesis by exploring whether 3 months or 6 months of anti-IL17A treatment will prevent relapses after medication has been discontinued in mild psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. 18 years of age or older
3. Chronic plaque-type psoriasis for at least 6 months
4. Negative PPD (negative chest w-ray if positive) or negative QuantiFERON-TB Gold
5. Have a PASI between 6 and 12 and Body Surface Area (BSA) affected by plaque-type psoriasis less than 10% at screening and baseline
6. Willing to wash off steroid creams and ultraviolet B light (UVB) therapy for 2 weeks prior to the baseline visit

Exclusion Criteria:

1. Has a nonplaque form of psoriasis (eg, erythrodermic, guttate, or pustular)
2. Has previously received Secukinumab or other biologics
3. History of Inflammatory Bowel Disease (IBD)
4. History of Rheumatoid Arthritis
5. Use of topical treatments for psoriasis, including steroids, vitamin D derivatives, vitamin A derivatives, salicylic acid, tar (except moisturizers) and/or ultraviolet A light (UVA)/UVB phototherapy within the last 2 weeks (if these have used them, the participant needs to wash off of them for at least 2 weeks after signing consent prior to baseline)
6. Is pregnant, nursing, or planning a pregnancy (both men and women) within 5 months following the last administration of study drug
7. Has recently received or is planning to receive a vaccination while on the study
8. HIV positive
9. Chronic untreated hepatitis C, positive hepatitis B surface antigen and acute hepatitis A infection
10. Known tuberculosis (TB) or evidence of TB infection. Subjects with a positive QuantiFERON; TB test or a positive purified protein derivate (PPD) skin test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active TB.
11. Any severe, progressive or uncontrolled medical condition at screening that in the judgment of the investigator prevents the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G Krueger, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller Univesity, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim J, Bissonnette R, Lee J, Correa da Rosa J, Suarez-Farinas M, Lowes MA, Krueger JG. The Spectrum of Mild to Severe Psoriasis Vulgaris Is Defined by a Common Activation of IL-17 Pathway Genes, but with Key Differences in Immune Regulatory Genes. J Invest Dermatol. 2016 Nov;136(11):2173-2182. doi: 10.1016/j.jid.2016.04.032. Epub 2016 May 13. PMID 27185339
- [Background] Kim J, Oh CH, Jeon J, Baek Y, Ahn J, Kim DJ, Lee HS, Correa da Rosa J, Suarez-Farinas M, Lowes MA, Krueger JG. Molecular Phenotyping Small (Asian) versus Large (Western) Plaque Psoriasis Shows Common Activation of IL-17 Pathway Genes but Different Regulatory Gene Sets. J Invest Dermatol. 2016 Jan;136(1):161-172. doi: 10.1038/JID.2015.378. PMID 26763436
- [Background] Kim J, Nadella P, Kim DJ, Brodmerkel C, Correa da Rosa J, Krueger JG, Suarez-Farinas M. Histological Stratification of Thick and Thin Plaque Psoriasis Explores Molecular Phenotypes with Clinical Implications. PLoS One. 2015 Jul 15;10(7):e0132454. doi: 10.1371/journal.pone.0132454. eCollection 2015. PMID 26176783
- [Background] Kim J, Krueger JG. The immunopathogenesis of psoriasis. Dermatol Clin. 2015 Jan;33(1):13-23. doi: 10.1016/j.det.2014.09.002. PMID 25412780

RESULTS

PARTICIPANT FLOW:
Groups:
- Secukinumab Only: 6 months of Secukinumab at a dose of 300 mg with injections administered once weekly at baseline and at weeks 1, 2, 3, and 4 and then every 4 weeks for 6 months of period.
  Secukinumab: Arms: Group 1 - Group 1 will receive Secukinumab at a dose of 300 mg with injections administered once weekly at baseline and at weeks 1, 2, 3, and 4 and then every 4 weeks for 6 months of period. In order to maintain the blind for the Group 2, Group 1 will receive placebo injections at weeks 13, 14, and 15. Group 1 will discontinue Secukinumab after 6 months of period being observed from week 25 to week 72 (48 weeks).
- Placebo Then Secukinumab: Placebo followed by Secukinumab. 3 months of placebo followed by 3 months of Secukinumab at a dose of 300 mg with injections administered once weekly at week 12 and at weeks 13, 14, 15, and 16 and then every 4 weeks for 3 months of period.
  Placebo followed by Secukinumab: Arms: Group 2 - Group 2 will receive placebo injections corresponding to the Group 1 regimen until week 8 in order to maintain a double-dummy design until week 12. From week 12, Group 2 will receive Secukinumab with injections administered once weekly at week 12 and at weeks 13, 14, 15, and 16 and then every 4 weeks for 3 months of period. Group 2 will discontinue Secukinumab after 6 months of period being observed from week 25 to week 72 (48 weeks).
Period: Overall Study
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [36.25 to 62.75] | 43 [40 to 57] | 44.0 [38.0 to 59.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
Psoriasis Area-Severity Index (PASI) [Median (Inter-Quartile Range); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
  units on a scale | 7.100 [6.100 to 9.450] | 8.900 [7.000 to 10.100] | 8.200 [6.100 to 9.950]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have 75% or More Reduction in [Psoriasis Area-and-severity Index Score (PASI)] (PASI75)
Description: The percentage of subjects who have a reduction of 75% or more from baseline in the Psoriasis Area and Severity Index (PASI) at week 12 (PASI 75). Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Time Frame: week 12
Population: One participant in Group 1 was not included in the data analysis due to a serious adverse event before the primary endpoint, unrelated to study medication or study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 11
Participants | 8 | 0

2. Secondary Outcome: Percentage of Subjects Who Have 90% or More Reduction in [Psoriasis Area-and-severity Index Score (PASI)] (PASI90)
Description: The percentage of subjects who have a reduction of 90% or more from baseline in the Psoriasis Area and Severity Index (PASI) at week 12 (PASI 90). Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 11
Participants | 7 | 0

3. Secondary Outcome: Percentage of Subjects Who Achieve a Physician Global Assessment (PGA) Score of 0 or 1 With at Least a 2-step Improvement From Baseline (PGA 0/1 Response Rate).
Description: Percentage of Subjects Who Achieve a Physician Global Assessment (PGA) score of 0 or 1 with at least a 2-step improvement from baseline (PGA 0/1 response rate). Physician Global Assessment (PGA) is a global assessment of all psoriasis lesions scored on a scale of 0-5, with 0 representing clear skin, 1 almost clear skin, and 5 representing severe psoriasis
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 11
Participants | 9 | 0

4. Secondary Outcome: Percentage of Subjects Who Experience Psoriasis Relapse
Description: The percentage of subjects who experience a psoriasis relapse at any time between week 24 and week 72. Psoriasis relapse is defined as loss of > 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at week 24. Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Time Frame: week 24 through week 72
Population: The overall number of participants analyzed is lower than the total enrollment for the study, because of loss to follow up during the observation period between week 24 and week 72. The loss to follow-up disabled the statistical analyses of the outcome measure data. There were various reasons for loss to follow-up including the negative impacts of COVID-19 to the participants during the observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 6 | 3
Participants | 3 | 2

5. Secondary Outcome: Percentage of Subjects Who Experience Severe Psoriasis Relapse
Description: The percentage of subjects who experience a severe psoriasis relapse at any time between week 24 and week 72. Severe psoriasis relapse is defined as loss of > 75% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at week 24. Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Time Frame: Observation Period: week 24 through week 72.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 6 | 3
Participants | 2 | 1

6. Secondary Outcome: Percentage of Subjects Who Experience Psoriasis Relapse After Psoriasis is Cleared
Description: The percentage of subjects who experience a psoriasis relapse at any time between week 24 and week 72 among the subjects whose psoriasis is cleared between week 0 and week 24. Psoriasis relapse is defined as loss of > 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at week 24. Psoriasis clearance is defined as the achievement of PASI100, which is a reduction of 100% from baseline in the Psoriasis Area and Severity Index (PASI) score. Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Time Frame: Observation Period: week 24 through week 72
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 4 | 1
Participants | 1 | 1

7. Secondary Outcome: Elapsed Time Until Relapse
Description: Elapsed time from week 24 until relapse occurs before week 72, measured in weeks.
Time Frame: week 24 until week 72
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 3 | 2
weeks | 24 [18 to 24] | 48 [48 to 48]

8. Secondary Outcome: Percentage of Subjects Who Have 100% Reduction in [Psoriasis Area-and-severity Index Score (PASI)] (PASI100)
Description: The percentage of subjects who have a reduction of 100% from baseline in the Psoriasis Area and Severity Index (PASI) score (PASI100) at week 12. Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 11
Participants | 4 | 0

9. Secondary Outcome: Frequency of Adverse Events
Description: Frequency of all Adverse Events (AEs) including Serious Adverse Events (SAEs) that occur during the whole trial including the observational period (AEs and SAEs include but not limited to comorbidities, such as hypertension, diabetes, and cardiovascular diseases).
Time Frame: week 0 through week 72
Measure: Number; unit: events
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 12 | 11
events | 22 | 13

10. Secondary Outcome: Frequency of Serious Adverse Events
Description: Frequency of Serious Adverse Events (SAEs) that occur during the whole trial including the observational period.
Time Frame: week 0 through week 72
Measure: Number; unit: events
Arm/Group | Secukinumab Only | Placebo Then Secukinumab
Number analyzed (Participants) | 12 | 11
events | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/11
Other Adverse Events (participants affected / at risk) | 10/12 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12) | Group 2 (N=11)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12) | Group 2 (N=11)
eye disorders- blepheritis (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
tooth infection (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 5 (5) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neoplasms benig, malignant and unspecified (incl cysts and polyps), other: breast cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin and subcutaneous tissue disorders, other: folliculitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03131570/Prot_SAP_000.pdf